CLINICAL TRIAL: NCT04194515
Title: Gut Microbiota and Bile Acids Mediate the Clinical Benefits of Metformin and YH1 in Patients With Treatment-naïve Type 2 Diabetes Mellitus: A Pilot Observational Study
Brief Title: Gut Microbiota and Bile Acids in Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901022A3C601
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2; Metformin; YH1
Keywords: Bile acid; Microbiota
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- YH1 group
  Interventions: Drug: YH1
- Metformin group
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: YH1 — YH1 treatment for one month
  Groups: YH1 group
Drug: metformin — metformin treatment for one month
  Groups: Metformin group

SUMMARY:
The investigators will evaluate the stool microbiota, serum and fecal bile acid composition, and changes in blood glucose and lipid profile before and after one month of metformin or YH1 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naïve male patients with type 2 diabetes;
2. Aged 20-65 years;
3. Body mass index (BMI) ≥ 24 kg/m2; 4.7 % ≤ glycated hemoglobin (HbA1c) < 9 %;

5.Low-density cholesterol (LDL-C) ≥ 130 mg/dl; 6.Expected to receive metformin 500 mg tid or YH1 6g tid for one month

Exclusion Criteria:

1. type 1,or other specific types of diabetes;
2. female;
3. history of oral hypoglycemic agents (OHAs) treatment or insulin therapy;
4. use of lipid-lowering drugs within the past six months;
5. serious gastrointestinal (GI) tract diseases, including peptic ulcers and GI tract bleeding;
6. hepatic insufficiency with ALT >72 U/L or renal insufficiency with an eGFR < 60 mL/min/1.73 m2;
7. history of stressful situations, including diabetic ketoacidosis, nonketotic hyperosmolar diabetic coma, infectious disease, or surgery in the previous month;
8. mental illness;
9. current smoking status, alcohol or drug abuse;
10. hemoglobin disease or chronic anemia;
11. underlying conditions that could lead to poor compliance;
12. severe organic diseases, including cancer, coronary heart disease, myocardial infarction or cerebrovascular disease;
13. continuous antibiotic or probiotics use for over 3 days within 3 months prior to enrollment;
14. continuous use of weight loss drug for over 1 month;
15. history of YH1 therapy, or Chinese medicine treatment within the past one month.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients and treatment-naïve male patients with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
bile acid profile | one month
  before and after YH1 or metformin treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided